CLINICAL TRIAL: NCT05789784
Title: Multicenter Prospective Study of Zimmer Biomet Mymobility Application on Reverse Total Shoulder Arthroplasty (RTSA) Outcomes
Brief Title: Study of Zimmer Biomet Mymobility Application on Reverse Total Shoulder Arthroplasty (RTSA) Outcomes
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Campbell Clinic (Other)
Collaborators: American Shoulder and Elbow Surgeons (Other)
Responsible Party: Principal Investigator, Tyler J. Brolin, Assistant Professor, Shoulder and Elbow Surgery, Co-director Shoulder and Sports Medicine Fellowship, Campbell Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 23-09443-FB
Record Dates: First submitted 2023-03-16; First posted 2023-03-29 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Reverse Total Shoulder Arthroplasty; Physical Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mymobility Physical Therapy (Experimental): The mymobility Physical Therapy cohort will complete an identical protocol to the Standard Office-based Physical Therapy cohort with one exception: the mymobility cohort's therapy for the entire duration of the protocol is administered at home through the mymobility application. This cohort initiates use of the mymobilty application one postoperative day 1. Exercises and restrictions are described in-depth in the Study Protocol document.
  Interventions: Other: mymobility Physical Therapy
- Standard Office-based Physical Therapy (Active Comparator): The Standard Office-based Physical Therapy cohort completes an identical protocol to the mymobility Physical Therapy cohort with one exception: rather than through use of the mymobility application, the Standard Office-based Physical Therapy cohort's protocol is administered through the traditional means of an exercise handout for postoperative day 1 through 2 weeks followed by formal office-based physical therapy for the duration of the protocol. Exercises and restrictions are described in-depth in the Study Protocol document.
  Interventions: Other: Standard Office-based Physical Therapy

INTERVENTIONS:
Other: mymobility Physical Therapy — Physical therapy protocol administered at home through the mymobility application.
  Arms: mymobility Physical Therapy
Other: Standard Office-based Physical Therapy — Physical Therapy protocol administered through exercise handouts and formal office-based therapy directed by physical therapist.
  Arms: Standard Office-based Physical Therapy

SUMMARY:
This is a trial comparing self-directed rehabilitation using the Zimmer Biomet mymobility digital platform versus standard office-based physical therapy after reverse shoulder replacement. The investigators hypothesize that there will be no difference in the postoperative outcomes between the mymobility cohort and the standard office-based physical therapy cohort.

DETAILED DESCRIPTION:
This is a prospective, multicenter, randomized controlled trial comparing a self-directed rehabilitation protocol using the Zimmer Biomet mymobility digital platform versus standard office based physical therapy protocol after reverse total shoulder arthroplasty.

Subjects will be randomly assigned to the Treatment Cohort (mymobility Physical Therapy) or the Control Cohort (Standard Office-based Physical Therapy). Randomization will occur following completion of a signed consent form. Each Participating Site will receive sealed, numbered randomization envelopes from the Lead Site.

The treatment cohort is mymobility PT. If the subject is randomized to this cohort, the Participating Site will assist the subject to download the mymobility mobile application (app) during the preoperative visit. The app has a video of each of the exercises to be completed per phase of the rehabilitation protocol beginning on postop day one.

The control cohort is Standard office PT. Home exercises begin on postoperative day one with office visits beginning after the 2 week postoperative visit.

Subject data will be collected through the 6-month postoperative visit.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older.
* Primary Reverse Total Shoulder Arthroplasty performed for diagnosis of cuff tear arthropathy (CTA), massive rotator cuff tears (mRCT), osteoarthritis (OA), or inflammatory arthritis (IA).
* Have a functioning smartphone model compatible with the mymobility platform.

Exclusion Criteria:

* Less than 18 years of age.
* Revision Reverse Total Shoulder Arthroplasty
* Concomitant tendon transfer
* Planned discharge to inpatient rehab facility, skilled nursing home, or use of home health therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-10-31 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
American Shoulder and Elbow Surgeons (ASES) Standardized Shoulder Assessment Score | 6 months
  The ASES Standardized Shoulder Assessment Score outputs a measurement of patient pain and function on a scale of 0 to 100, with 0 being the greatest pain and no function and 100 being no pain and perfect function.

CONTACTS AND LOCATIONS:
Overall Officials: Tyler J Brolin, MD, Principal Investigator — Campbell Clinic
Locations (4):
- United States (4):
  - Atlantis Orthopedics, Palm Beach Gardens, Florida
  - Ohio State University Medical Center, Columbus, Ohio
  - Rothman Orthopaedic Institute, Philadelphia, Pennsylvania
  - Campbell Clinic, Germantown, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wagner ER, Farley KX, Higgins I, Wilson JM, Daly CA, Gottschalk MB. The incidence of shoulder arthroplasty: rise and future projections compared with hip and knee arthroplasty. J Shoulder Elbow Surg. 2020 Dec;29(12):2601-2609. doi: 10.1016/j.jse.2020.03.049. Epub 2020 Jun 9. PMID 33190759
- [Background] Crawford DA, Lombardi AV Jr, Berend KR, Huddleston JI 3rd, Peters CL, DeHaan A, Zimmerman EK, Duwelius PJ. Early outcomes of primary total hip arthroplasty with use of a smartphone-based care platform: a prospective randomized controlled trial. Bone Joint J. 2021 Jul;103-B(7 Supple B):91-97. doi: 10.1302/0301-620X.103B7.BJJ-2020-2402.R1. PMID 34192907
- [Background] Crawford DA, Duwelius PJ, Sneller MA, Morris MJ, Hurst JM, Berend KR, Lombardi AV. 2021 Mark Coventry Award: Use of a smartphone-based care platform after primary partial and total knee arthroplasty: a prospective randomized controlled trial. Bone Joint J. 2021 Jun;103-B(6 Supple A):3-12. doi: 10.1302/0301-620X.103B6.BJJ-2020-2352.R1. PMID 34053272
- [Background] Yayac M, Moltz R, Pivec R, Lonner JH, Courtney PM, Austin MS. Formal Physical Therapy Following Total Hip and Knee Arthroplasty Incurs Additional Cost Without Improving Outcomes. J Arthroplasty. 2020 Oct;35(10):2779-2785. doi: 10.1016/j.arth.2020.04.023. Epub 2020 Apr 18. PMID 32674941
- [Background] Simovitch RW, Friedman RJ, Cheung EV, Flurin PH, Wright T, Zuckerman JD, Roche C. Rate of Improvement in Clinical Outcomes with Anatomic and Reverse Total Shoulder Arthroplasty. J Bone Joint Surg Am. 2017 Nov 1;99(21):1801-1811. doi: 10.2106/JBJS.16.01387. PMID 29088034
- [Background] Kolin DA, Moverman MA, Pagani NR, Puzzitiello RN, Dubin J, Menendez ME, Jawa A, Kirsch JM. Substantial Inconsistency and Variability Exists Among Minimum Clinically Important Differences for Shoulder Arthroplasty Outcomes: A Systematic Review. Clin Orthop Relat Res. 2022 Jul 1;480(7):1371-1383. doi: 10.1097/CORR.0000000000002164. Epub 2022 Mar 17. PMID 35302970